CLINICAL TRIAL: NCT00563160
Title: Phase II Study of the Response Rate of Induction Chemotherapy With Gemcitabine and Carboplatin for Operable Non-small Cell Lung Cancer Before Surgery
Brief Title: Study of Efficacy of Induction Chemotherapy With Gemcitabine and Carboplatin for Operable Non-small-cell Lung Cancer Before Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (193-h)in QE/EC/I; HARECCTR0500015; 000904; B9E-IH-O333
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Lung Neoplasms
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Carboplatin; Surgical Procedures, Operative

INTERVENTIONS:
Drug: gemcitabine, carboplatin
Procedure: surgery

SUMMARY:
To study the activity of chemotherapy with Gemzar-carboplatin in the preoperative setting for operable stages of non-small-cell lung cancer and to identify novel molecular markers correlated with chemosensitivity and prognosis

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven, newly diagnosed primary bronchogenic non-small cell lung cancer
* Measurable or evaluable tumour on chest X-ray or CT scan.
* No multiple ipsilateral or contralateral parenchymal tumours
* Stage I(exceptT1N0),II,IIIa disease as shown by PET-CT

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05; Study Completion 2007-02 (Estimated)

PRIMARY OUTCOMES:
pathological response rate | 12 months

SECONDARY OUTCOMES:
progression-free survival | 18 months
overall survival | 18 months
quality of life measurements | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Siu Kie Au, Dr, Principal Investigator — Department of Clinical Oncology, Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, China